CLINICAL TRIAL: NCT01870687
Title: Prospective, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Randomized Clinical Trial to Proof Efficacy and Safety of 20 mg (2 Tablets of 10 mg) VAC BNO 1095 FCT in Patients Suffering From Cyclic Mastodynia and PMS
Brief Title: Efficacy and Safety of 20 mg (2 Tablets of 10mg)VAC BNO 1095 FCT on Cyclic Mastodynia and PMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-AG-E-4; 2012-005042-37
Record Dates: First submitted 2013-05-16; First posted 2013-06-06 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Premenstrual Syndrome; Mastodynia
Keywords: vitex agnus castus; clinical trial; cyclic mastodynia; PMS; prospective
MeSH Terms: conditions — Premenstrual Syndrome; Mastodynia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAC BNO 1095 2x10 mg FCT (Experimental): VAC BNO 1095 2x10 mg FCT 2 tablets of verum in the morning, oral, 3 months treatment
  Interventions: Drug: 20mg VAC BNO 1095 FCT
- Placebo (Placebo Comparator): 2 tablets in the morning, oral, 3 months treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20mg VAC BNO 1095 FCT
  Arms: VAC BNO 1095 2x10 mg FCT
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to proof the efficacy and safety of 20 mg (2 tablets of 10 mg) VAC BNO 1095 film-coated tablets in patients suffering from cyclic mastodynia and PMS (pre menstrual syndrome).

DETAILED DESCRIPTION:
The study consists of a 2-cycle run-in period, followed by 3 cycles of treatment. After first screening at S-2 further visits are scheduled after the end of each of the first and second run-in cycle, and after the first, second and third treatment cycle, respectively.

At least 220 patients should be eligible for randomisation, 110 to each treatment group, of which 160 (80 per group) will be available for data evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 to 45 Y with a history of cyclic mastodynia and PMS
* Stable cycle duration of 25 to 35 days.
* Subject is reporting at least one moderate or severe physical PMS symptom moderate and one psychic symptom, using the COPE symptom list
* Subject is reporting symptoms of a total score of at least 15 in the late luteal phase of the preceding cycle, using the COPE symptom list
* In both run-in cycles: Confirmation of cyclic mastodynia based on daily recordings of patient diary (VAS and COPE data)
* Subject provides a negative pregnancy test at study start and is willing to use a hormone-free medically acknowledged contraception methods with a PEARL-index < 1 % from enrolment
* Unsuspicious breast USG/mammogram not older than 12 months ruling out signs of malignancy

Exclusion Criteria:

* Hypersensitivity to the active substance or to the excipients of the IMP
* Proof of PMDD according to DSM IV criteria as defined by APA
* Intake of any of the following medications before treatment start and within 6 months prior to screening visit:

  * hypothalamic hormones
  * injectable contraceptives: 3-month injection
* Intake of any of the following medications (including herbal or homeopathic drugs) before treatment start and within 3 months prior to screening visit:

  * any treatment for mastodynia or premenstrual complaints
  * sexual hormones, combinations and inhibitors
  * pituitary hormones and their inhibitors
  * dopamine-agonists and dopamine-antagonists
  * neuroleptics, antidepressants (including serotonin- and serotonin-norepinephrine-reuptake-inhibitors)
  * prolactin-inhibitors or prolactin stimulating preparations
  * drug abuse or continuous intake of NSAIDs or any other analgetics including antirheumatics (up to 2 tablets of paracetamol 500 mg or equivalent per week are allowed)
  * spironolactone
  * gonadotrophin inhibitors
  * diuretics
  * danazol
  * psychotropic agents
* Any psychiatric treatment before treatment start and within 12 months prior to screening visit
* Medical history or presence of any of the following medical conditions/ diseases before treatment start:

  * Uncontrolled diabetes mellitus: Patients with known diabetes mellitus, who have a glycosylated haemoglobin (HbA1c) ≥ 7% as assessed at visit S-1
  * Uncontrolled hypertension: Patients with a diastolic blood pressure >90mmHg at visit S-2
  * Known cardiac insufficiency, coronary heart disease, valvular heart disease, cardiac arrhythmia, QT interval prolongation or other severe cardiac disease at visit S-2
  * Known clinically significant organ or systemic diseases or any other relevant medical condition such that in the opinion of the investigator, the significance of the disease or condition will compromise the subject's participation in the study
  * Known hyperprolactinemia (serum prolactin basal > 50 ng/ml or > 1050 mlU/L)
  * Known hypo-/hyperthyreosis
  * Known hypo-/hyperparathyroidism
  * Known pituitary tumor including prolactinoma
  * Known chronic kidney disease
  * Known gastrointestinal, or liver diseases, such as:

    i. active peptic gastric ulcer ii. malabsorption iii. hepatitis
  * endometriosis
  * breast cancer, fibroadenoma, intraductal papilloma or other malignancy within the last 10 years
  * suspicious non-verified finding on any breast ultrasound or mammograms in the past
  * galactorrhea of degree II or III
  * purulent or bloody nipple discharge
  * refractory and/or unverified breast skin- or nipple/areola lesions
  * pregnancy, lactation
  * wish for pregnancy
  * any surgery planned to take place during the trial including breast cyst puncture
* Values of safety laboratory parameters outside normal ranges and clinically relevant as assessed by the investigator at S-1
* At screening:TSH > 2.5 mU/L
* Patients who have difficulties in understanding the language in which the patient information is given
* Patients who are members of the staff of the study centre, staff of the sponsor or CRO, the investigator herself or close relatives of the investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum severity of cyclic breast pain | after 3 months treatment under Investigational Medicinal Product (IMP).
  Maximum severity of cyclic breast pain after 3 months treatment under Investigational Medicinal Product (IMP). The severity of cyclic breast pain will be self-assessed by the patient on a Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Severity of cyclic breast pain and PMS symptoms | After 1, 2 and 3 months of treatment
  * Maximum severity of cyclic breast pain after 1 and 2 months treatment, respectively. The severity of cyclic breast pain will be self-assessed by the patient on a VAS
  * Average severity of cyclic mastodynia, determined in the late luteal phase of each of the treatment cycles.
  * Intensity of PMS assessed by means of a PMS diary (COPE = calendar of premenstrual experiences) during each of the treatment cycles
  * Overall assessments of efficacy on cyclic mastodynia and PMS by patient and investigator at study end by a score ranging from 1 to 5
  * Subgroup analysis: A. Patients with the waist circumference ≤ 90 cm B. Patients with the waist circumference > 90 cm. For both subgroups A. and B.: Maximum severity of cyclic breast pain after 3 months treatment under IMP. The severity of cyclic breast pain will be self-assessed by the patient on a VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Witek, MD PhD Prof., Study Chair; Hannes Herold, Dr. med., Study Chair
Locations (1):
- Private Doctor's office - Dr. Hannes Herold, Munich, Bavaria, Germany